CLINICAL TRIAL: NCT01560208
Title: The Asia Cornea Society Infectious Keratitis Study
Acronym: ACSIKS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asia Cornea Society (Other)
Collaborators: Singapore Clinical Research Institute (Other)
Responsible Party: Principal Investigator, Prof Donald TH Tan, Principal Investigator and Chairman, ACSIKS Council, Asia Cornea Society
Other Study IDs: ACSIKS
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Corneal Ulcer
Keywords: infectious keratitis; infective keratitis; prospective multicentre study; Asia
MeSH Terms: conditions — Corneal Ulcer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Positive bacterial and fungal growth obtained from the cornea samples of ACSIKS patients will be retained and stored.
Oversight: Data Monitoring Committee: No

SUMMARY:
Corneal diseases are a major cause of blindness worldwide, and corneal infections are a substantial cause of blindness in Asia. The aim of the Asia Cornea Society Infectious Keratitis Study (ACSIKS) is to study infectious keratitis (corneal infections) in Asian countries, so as to improve strategies for prevention and treatment, and to reduce the burden of blindness in Asia.

The first phase of ACSIKS is an 18-month observational study involving 11 eye hospitals in 8 Asian countries; these hospitals manage more than 6700 cases of corneal infections every year. From the first quarter of 2012, all patients with a corneal infection will be recruited and a standard ACSIKS protocol will be applied; this protocol includes the use of a common set of study forms and a suggested panel of microbiological examinations. However, each centre will be continue to treat their patients with the anti-infective therapy standard for their centre. Data will be recorded for each patient for a period of six months, including their medical and surgical management, the final clinical outcome and vision.

Bacterial and fungal growths from patients will also be stored for further research during a second phase of ACSIKS. These studies will focus on evaluating the resistance of the most common bacterial infections to the current available antibiotics, performing DNA testing to compare our strains with bacterial infections in the West, and to developing new diagnostic tests and anti-infective therapies tailored to corneal infections in Asia.

DETAILED DESCRIPTION:
Summary of the ACSIKS Clinical Protocol:

All patients with an initial clinical diagnosis of infectious keratitis will be referred by the attending ophthalmologist-in-charge to an ACSIKS co-investigator or trial coordinator for recruitment into the study. Patients will be enrolled in the study after study informed consent is obtained and a trained interviewer will administer a standardized ACSIKS Clinical Case Report Form to each recruited subject. Information that will be documented would include the demographic profile (e.g. age, gender, ethnic group, occupation, etc), risk factors for infectious keratitis, presenting symptoms and prior treatment.

Patients who are contact lens wearers will also complete a separate contact lens questionnaire, with specific questions on duration of contact lens wear, type of contact lens and solutions used, lens wear schedule and habits, and adherence to lens care practices.

All patients will undergo a thorough ocular examination by the ophthalmologist-in-charge or an ACSIKS co-investigator, and details of the infectious keratitis and associated findings documented on the ACSIKS Clinical CRF. With the approval of the ophthalmologist-in-charge, corneal scrapings will then be collected as per the ACSIKS Microbiological Protocol. Each study subject will consequently still be managed by the ophthalmologist-in-charge according to his/her current clinical approach, with appropriate medical or surgical treatment carried out in accordance with the practice patterns and standards of his/her institution, and no attempt to deviate from current treatment practices.

Regular chart reviews will be performed by ACSIKS trial coordinators for the six months duration of the subjects' involvement to document the initial differential diagnoses and medical treatment, the microbiological results, and any changes to the diagnosis and treatment. The last consultation with the ophthalmologist-in-charge during that six month-period will be taken as the final study review.

Summary of the ACSIKS Microbiological Protocol:

At the discretion of the ophthalmologist-in-charge, corneal scrapings will be collected based on a list of investigations suggested by the ACSIKS Group.

All microbiological specimens will be incubated, interpreted and reported according to agreed upon common standards, regardless of the number of colonies present. Bacterial organisms will also be tested using standardized antibiograms agreed upon by microbiologists from the various participating institutions. Results of any and all microbiological testing will be collected and recorded into the ACSIKS Microbiological Case Report Form.

If these samples do yield a positive growth of either fungal or bacterial organisms (or both), the causative organisms cultured will be sub-cultured and stored at each site's ACSIKS freezer, for subsequent transport to the ACSIKS Central Repository in Singapore for use in future microbial studies under Phase 2 of the ACSIKS project.

ELIGIBILITY:
Inclusion Criteria:

* all patients presenting to an ACSIKS site during the study period with an initial diagnosis of infectious keratitis in one or both eyes

Exclusion Criteria:

* patients who are cognitively impaired or otherwise unable to give direct informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ACSIKS will recruit all patients with infectious keratitis from 11 Study Centres in eight different countries (India, China, Japan, South Korea, Taiwan, Thailand, the Philippines and Singapore), each evaluating all cases of infectious keratitis presenting over a 12 month period.
  There will be a total of 11 Study Centres¸ with India, China and Japan each having 2 separate study centres. Some Study Centres will also be responsible for coordinating cases accrued from affiliated hospitals ("Participating Institutions").
Sampling Method: Probability Sample
Enrollment: 6750 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Resolution of infectious keratitis | 6 months from enrollment
  Resolution of the infectious keratitis occurs when the infiltrate clears, epithelium heals over, and inflammation subsides.

SECONDARY OUTCOMES:
Number of acute surgical interventions required. | 6 months from enrollment
  Any form of surgery performed during the acute stage of the infection. The number and type of surgery performed and the surgical outcomes will be captured.
Visual acuity outcome of management. | 6 months from enrollment
  Visual acuity will be documented. Reasons for poor visual acuity (less than 6/18 or 0.3) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Donald TH Tan, FRCS(G), Principal Investigator — Singapore National Eye Centre, Singapore Eye Research Institute, National University Hospital
Locations (11):
- China (2):
  - Shandong Eye Institute, Qingdao
  - Xiamen Eye Center, Xiamen
- India (2):
  - L.V.Prasad Eye Institute, Hyderabad, Andhra Pradesh
  - Aravind Eye Hospital, Madurai, Tamil Nadu
- Japan (2):
  - Department of Ophthalmology, Faculty of Medicine, Osaka University Graduate School of Medicine Hospital, Osaka
  - Department of Ophthalmology, Tottori University Hospital, Tottori
- Department of Ophthalmology and Visual Sciences, Philippine General Hospital, Manila, Philippines
- Singapore Eye Research Institute, Singapore, Singapore
- Department of Opthalmology & Visual Science, The Catholic University of Korea, Seoul St. Mary's Eye Institute, Seoul, South Korea
- Department of Opthalmology, National Taiwan University Hospital, Taipei, Taiwan
- Department of Ophthalmology, Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok, Thailand